CLINICAL TRIAL: NCT03670160
Title: Clonidine Versus Phenobarbital as Adjunctive Therapy for Neonatal Abstinence Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tennessee Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHS-OB-0001
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Phenobarbital; Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenobarbital (Active Comparator): Phenobarbital loading dose 20mg/kg in 2 divided doses, then 5 mg/kg/day divided every 12 hours. Phenobarbital continued throughout the infants hospitalization.
  Interventions: Drug: Phenobarbital
- Clonidine (Active Comparator): Clonidine 5 mcg/kg/day divided every 3 hours. Clonidine will be continued to achieve control of NAS symptoms. Clonidine may be weaned after successful discontinuation of oral morphine sulfate. Infants will not be discharged on clonidine.
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Phenobarbital — Phenobarbital loading dose 20 mg/kg in 2 divided doses, then 5 mg/kg/day divided every 12 hours. Phenobarbital dose will be adjusted to obtain desired trough of 25 to 30 mcg/mL. Levels will be obtained on Day 6 then weekly thereafter. Phenobarbital will be tapered over 4 weeks upon discharge from the hospital. The standardized taper is based the patient specific dose at the time of discharge.
  Arms: Phenobarbital
Drug: Clonidine — Clonidine 5 mcg/kg/day divided every 3 hours. Clonidine will be increased by 1.5 mcg/kg/day to achieve control of NAS symptoms based upon standardized scoring for neonatal abstinence syndrome. Clonidine will be weaned by 25% every 24 hours after successful discontinuation of oral morphine sulfate. Infants will not be discharged on clonidine.
  Arms: Clonidine

SUMMARY:
The purpose of this study is to compare clonidine versus phenobarbital as adjunctive therapy in those infants who have failed monotherapy with morphine sulfate for neonatal abstinence syndrome (NAS).

ELIGIBILITY:
Inclusion Criteria:

* Infants greater than or equal to 35 weeks gestation age
* Admitted to the neonatal intensive care unit
* Failed monotherapy with morphine sulfate therapy

Exclusion Criteria:

* Neonatal abstinence syndrome due to iatrogenic causes
* Unable to take oral medications at any point during their treatment
* Infants in the custody of the Department of Child Protective Services with no legal guardian identified at the time of enrollment

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Brusseau, PharmD, Principal Investigator — University of Tennessee Medical Center
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phenobarbital | Clonidine
Started | 11 | 14
Completed | 11 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenobarbital | Clonidine | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 14 | 25
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 38 (1) | 38.6 (1.6) | 38.3 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 14 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 14 | 25
Appearance, Pulse, Grimace, Activity, and Respiration - APGAR scale [Mean (Standard Deviation); unit: units on a scale] — The APGAR scale assigns a numerical value of 0-10 (0-2 to each of the 5 items with 2 being the best). A combined score of 7 or higher is considered normal.
  units on a scale | 6.7 (2.1) | 7.8 (0.9) | 7.3 (1.4)
Birth weight, grams [Mean (Standard Deviation); unit: Grams] | 3173 (588) | 3141 (519) | 3155 (549)

OUTCOME MEASURES:

1. Primary Outcome: Time From Initiation of Adjunctive Therapy Until Hospital Discharge
Description: Number of days from initiation of adjunctive therapy until hospital discharge
Time Frame: From date of randomization until hospital discharge, up to 4 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phenobarbital | Clonidine
Number analyzed (Participants) | 11 | 14
Days | 20 (12.6) | 33.8 (14.3)

2. Secondary Outcome: Length of Stay
Description: Number of days of hospital admission
Time Frame: From date of randomization until hospital discharge, up to 4 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phenobarbital | Clonidine
Number analyzed (Participants) | 11 | 14
Days | 31 (9.96) | 41.78 (10.94)

3. Secondary Outcome: Length of Oral Morphine Sulfate Therapy
Description: Number of days of oral morphine sulfate therapy
Time Frame: From date of randomization until hospital discharge, up to 4 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phenobarbital | Clonidine
Number analyzed (Participants) | 11 | 14
Days | 25.45 (6.95) | 34.36 (10.18)

4. Secondary Outcome: Number of Patients Requiring Triple Therapy
Description: Number of patients requiring a third agent to control withdrawal symptoms
Time Frame: From date of randomization until hospital discharge, up to 4 months
Measure: Number; unit: participants
Arm/Group | Phenobarbital | Clonidine
Number analyzed (Participants) | 11 | 14
participants | 4 | 10

5. Secondary Outcome: Readmission Rate
Description: Number of patients readmitted to the hospital within 30 days of hospital discharge or discontinuation of phenobarbital.
Time Frame: From date of randomization until 30 days after hospital discharge or discontinuation of phenobarbital, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phenobarbital | Clonidine
Number analyzed (Participants) | 11 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Phenobarbital | Clonidine
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 0/11 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenobarbital (N=11) | Clonidine (N=14)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2) — Clonidine dose held - 2 infants developed hypotension requiring additional clonidine weaning to resolve.
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) — Clonidine dose held. 1 infant experienced rebound hypertension which resolved with no clonidine wean adjustment to resolve.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT03670160/Prot_SAP_000.pdf